CLINICAL TRIAL: NCT01623245
Title: Prevalence of Transthyretin Amyloidosis in Hypertrophic Cardiomyopathy
Acronym: Amylo
Status: Completed | Type: Observational
Sponsor: Thibaud Damy (Other)
Responsible Party: Sponsor-Investigator, Thibaud Damy, Assistant Professor, French Cardiology Society
Organization: French Cardiology Society (Other)
Other Study IDs: 11714
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Amyloidosis; Amyloidosis in Transthyretin (TTR); Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL of whole blood in EDTA tube
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypertrophic Cardiomyopathy: In the population of Hypertrophic Cardiomyopathy patients, patients suffering from a cardiac amyloidosis

SUMMARY:
Cardiac amyloidosis are related to the accumulation of fibrillar proteins in the extracellular leading to disruption of the cardiac tissue architecture. Amyloidosis in transthyretin (TTR) are the most common hereditary amyloidosis but remain poorly studied at heart. This is serious and deadly. The prevalence of TTR amyloidosis is probably underestimated in hypertrophic cardiomyopathy (HCM) often of unknown etiology because of the lack of systematic implementation of myocardial biopsy because of their side effects.

DETAILED DESCRIPTION:
A systematic screening of TTR mutations within the MHC would diagnose cardiac amyloidosis in TTR and improve the care of patients and their families.

The detection of this disease is important because this disease is fatal and a new treatment to prevent the accumulation of TTR is now available (Tafamidis). This drug has proved effective in stabilizing neurological damage.

Depending on the number of patient with cardiac amyloidosis in TTR detected, the prospect will begin a clinical trial to test the effectiveness of a new treatment to prevent the increase in mass of the left ventricle wall objectified resonance nuclear Magnetic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiomyopathy defined by an ultrasound thickness of the left ventricle >= 13 mm if familial form or >= 15 mm if sporadic form.
* Patients with a signed consent authorizing the specific blood test for genetic sequencing to look for abnormal TTR gene

Exclusion Criteria:

* Patients with a diagnosis of cardiomyopathy already determined or related already diagnosed.
* Significant aortic stenosis (≤ 1 cm ²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is that of patients with hypertrophic cardiomyopathy in France whose origin has not yet been determined.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of ATTRm mutations | 1 day
  Number of ATTRm mutations detected in a large population of patients with HCM.

SECONDARY OUTCOMES:
Genotype and clinical factors | 1 day
  Identify clinical factors associated with biological and echocardiographic different HCM genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud DAMY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Christoph DC, Boese D, Johnson KT, Schlosser TW, Hunold P, Baba HA, Erbel R, Philipp S. Heart failure and cardiac involvement as isolated manifestation of familial form of transthyretin amyloidosis resulting from Val30Met mutation with no clinical signs of polyneuropathy. Circ Heart Fail. 2009 Sep;2(5):512-5. doi: 10.1161/CIRCHEARTFAILURE.109.853697. No abstract available. PMID 19808383
- [Background] Merlini G, Bellotti V. Molecular mechanisms of amyloidosis. N Engl J Med. 2003 Aug 7;349(6):583-96. doi: 10.1056/NEJMra023144. No abstract available. PMID 12904524
- [Background] Morner S, Hellman U, Suhr OB, Kazzam E, Waldenstrom A. Amyloid heart disease mimicking hypertrophic cardiomyopathy. J Intern Med. 2005 Sep;258(3):225-30. doi: 10.1111/j.1365-2796.2005.01522.x. PMID 16115295
- [Background] Jacobson DR, Pastore RD, Yaghoubian R, Kane I, Gallo G, Buck FS, Buxbaum JN. Variant-sequence transthyretin (isoleucine 122) in late-onset cardiac amyloidosis in black Americans. N Engl J Med. 1997 Feb 13;336(7):466-73. doi: 10.1056/NEJM199702133360703. PMID 9017939
- [Background] Plante-Bordeneuve V, Ferreira A, Lalu T, Zaros C, Lacroix C, Adams D, Said G. Diagnostic pitfalls in sporadic transthyretin familial amyloid polyneuropathy (TTR-FAP). Neurology. 2007 Aug 14;69(7):693-8. doi: 10.1212/01.wnl.0000267338.45673.f4. PMID 17698792
- [Background] Plante-Bordeneuve V. [The diagnosis and management of familial amyloid polyneuropathy]. Rev Neurol (Paris). 2006 Nov;162(11):1138-46. doi: 10.1016/s0035-3787(06)75130-x. French. PMID 17086153
- [Background] Rapezzi C, Merlini G, Quarta CC, Riva L, Longhi S, Leone O, Salvi F, Ciliberti P, Pastorelli F, Biagini E, Coccolo F, Cooke RM, Bacchi-Reggiani L, Sangiorgi D, Ferlini A, Cavo M, Zamagni E, Fonte ML, Palladini G, Salinaro F, Musca F, Obici L, Branzi A, Perlini S. Systemic cardiac amyloidoses: disease profiles and clinical courses of the 3 main types. Circulation. 2009 Sep 29;120(13):1203-12. doi: 10.1161/CIRCULATIONAHA.108.843334. Epub 2009 Sep 14. PMID 19752327
- [Background] Said G, Plante-Bordeneuve V. Familial amyloid polyneuropathy: a clinico-pathologic study. J Neurol Sci. 2009 Sep 15;284(1-2):149-54. doi: 10.1016/j.jns.2009.05.001. Epub 2009 May 24. PMID 19467548
- [Background] Saraiva MJ. Sporadic cases of hereditary systemic amyloidosis. N Engl J Med. 2002 Jun 6;346(23):1818-9. doi: 10.1056/NEJM200206063462312. No abstract available. PMID 12050344